CLINICAL TRIAL: NCT05241743
Title: Examining the Relationship Between Cervical Hypolordosis and Pain, Phone Addiction, and Nomophobia in Young Adults
Brief Title: The Relationship Between Cervical Hypolordosis and Pain, Phone Addiction, and Nomophobia
Status: Completed | Type: Observational
Sponsor: University of Beykent (Other)
Collaborators: Beylikduzu State Hospital (Other); Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Yasemin Şahbaz, doctoral lecturer, University of Beykent
Other Study IDs: UBeykent-1
Record Dates: First submitted 2021-11-01; First posted 2022-02-16 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Neck Pain
Keywords: neck pain; Nomophobia; phone addiction
MeSH Terms: conditions — Neck Pain | interventions — X-Rays

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: radiological examination, pain, nomophobia, phone addiction — 120 patients who applied to the clinic with the complaint of neck pain and were diagnosed with cervical hypolordosis by radiological examination will be included in the study. After giving the necessary verbal and written information about the study, a link will be sent to the phones of the patients whose informed consent was obtained. Patients will access evaluation questions and survey questions via this link. Personal information with the Sociodemographic Data Form prepared by us; pain severity by Visual Analogue Scale (VAS); phone addiction level with the Smartphone Addiction Questionnaire (Young Population); nomophobia levels will be evaluated with the Nomophobia Scale.

SUMMARY:
The aim of this study is to reveal the relationship between the degree of neck straightening and pain, phone addiction and nomophobia in young adult patients who applied to the clinic with the complaint of neck pain and were diagnosed with neck straightening as a result of radiological examinations.

120 patients who applied to the clinic with the complaint of neck pain and were diagnosed with cervical hypolordosis by radiological examination will be included in the study. After giving the necessary verbal and written information about the study, a link will be sent to the phones of the patients whose informed consent was obtained. Patients will access evaluation questions and survey questions via this link. Personal information with the Sociodemographic Data Form prepared by us; pain severity by Visual Analogue Scale (VAS); phone addiction level with the Smartphone Addiction Questionnaire (Young Population); nomophobia levels will be evaluated with the Nomophobia Scale.

DETAILED DESCRIPTION:
Indication or complications Patients between the ages of 18-35, diagnosed with neck flattening and who agreed to participate in the study will be included in the study. Patients under the age of 18 and older than 35, who cannot cooperate verbally and/or auditory, and who cannot cooperate psychologically and/or perceptually will be excluded from the study.

120 patients who applied to the clinic with the complaint of neck pain and were diagnosed with cervical hypolordosis by radiological examination will be included in the study. After giving the necessary verbal and written information about the study, a link will be sent to the phones of the patients whose informed consent was obtained. Patients will access evaluation questions and survey questions via this link. Personal information with the Sociodemographic Data Form prepared by us; pain severity by Visual Analogue Scale (VAS); phone addiction level with the Smartphone Addiction Questionnaire (Young Population); nomophobia levels will be evaluated with the Nomophobia Scale.

Sociodemographic Data Form: With the form, participants' name, surname, gender, age, height, weight, education status, marital status, smoking, alcohol, exercise habits, average daily sleep and smartphone usage time, screen usage time in the last 7 days, how many years smart phone usage information and contact information will be recorded.

Visual Analog Scale (VAS): participants are asked to select the point where they feel pain on a 10-centimeter (cm) horizontal line. 0 - no pain, 10 - unbearable pain. Pain conditions are evaluated separately at night, during activity and at rest.

Smartphone Addiction Questionnaire (Young Population): The scale consists of 33 questions and 7 sub-parameters. Sub-parameters Functioning Impairment, Withdrawal Symptom, Positive Expectation, Virtual Directed Relationship, Overuse, Social Network Addiction, and Physical are symptoms. As the score increases, the level of addiction increases. Nomophobia Scale: It has 20 items and 4 dimensions in total. These four dimensions, in order, are not being online, losing communication, not feeling comfortable, and not being able to access information. Each of the 20 questions in the 5-point Likert-type scale is scored by the participants as 1 point-strongly disagree, 7 points-strongly agree. If the total score is 20, it is graded as no nomophobia, 21-59 as mild nomophobia, 60-99 as moderate nomophobia, and 100-140 as extreme nomophobia.

Statistical analysis SPSS version 25 will be used in the analysis of the data. It will be evaluated whether the data are suitable for normal distribution. Descriptive statistics will be shown as mean ± standard deviation for variables with normal distribution, and median (min - max) for variables with non-normal distribution. Correlation tests will be used to check whether there is a relationship between the data.

For the relationship between independent variables, Spearman Correlation test or Pearson Correlation analysis will be performed according to the normal distribution and the level of significance will be accepted as p<0.05. If the correlation coefficient is r<0.2, it will be interpreted as very weak correlation or no correlation, between 0.2-0.4 as weak correlation, between 0.4-0.6 as moderate correlation, between 0.6-0.8 as high correlation and 0.8> as very high correlation.

Chronic neck pain is one of the most common musculoskeletal disorders. The cervical region contains many structures that can cause pain when damaged, such as muscles, ligaments, vertebrae, facet joints, intervertebral discs, spinal nerves. In addition, being the most mobile region of the vertebral column makes the cervical region vulnerable to possible traumas.

In the literature, it has been shown that long-term and repeated use of a smartphone while the neck is flexed causes neck pain. When using a smartphone, the device is usually held below eye level, one or both hands grasp the device, and the thumb is actively used to tap the screen and switch between apps. Prolonged protraction and flexion posture of the neck causes a spatial change between the spine and the line of gravity, causing overload in the muscles and connective tissues, leading to many problems such as discomfort, pain, reduction in cervical lordosis in smartphone users.

Technological developments in the last year have led to a significant increase in the use of mobile technology. According to the Household Information Technologies Usage Survey of the Turkish Statistical Institute, it was revealed that 96.9% of the households have mobile phones and smart phones in 2016. Especially the easy portability of smart phones, the increase in internet networks, and the easy access to information and entertainment content have increased the usage rates even more. Along with the Covid-19 Pandemic, young people, like all individuals in the society, had to stay away from their school, work and social circles within the scope of quarantine measures and have to stay at home. The use of on-line methods has increased in education and training activities, in the working system of many workplaces, in communication with family relatives and social environment. Whether this level of use has reached the level of addiction should be investigated. In addition to all these, the investigators observe that neck pain complaints increase due to the decrease in physical activity, the increase in the time spent with a smartphone, and the lack of attention to ergonomic principles during smartphone use. As far as the investigators know, there is no study in the literature examining the relationship between neck straightening, pain, phone addiction and nomophobia. Therefore, the investigators think that study will contribute to the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-35
* Diagnosed with neck flattening
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients under the age of 18 and older than 35,
* Who cannot cooperate verbally and/or auditory,
* Who cannot cooperate psychologically and/or perceptually

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who applied to the Department of Orthopedics and Traumatology of Beylikdüzü State Hospital with the complaint of neck pain and were diagnosed with cervical hypolordosis by radiological examination.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | through study completion, an average of 1 year
  Participants are asked to select the point where they feel their pain on a 10-centimeter (cm) horizontal line. 0 - no pain, 10 - unbearable pain. Pain conditions are evaluated separately at night, during activity and at rest.
Nomophobia | through study completion, an average of 1 year
  It has 20 items and 4 dimensions in total. These four dimensions, in order, are not being online, losing communication, not feeling comfortable, and not being able to access information. Each of the 20 questions in the 5-point Likert-type scale is scored by the participants as 1 point - strongly disagree, 7 points - strongly agree. If the total score is 20, it is graded as no nomophobia, 21-59 as mild nomophobia, 60-99 as moderate nomophobia, 100-140 as extreme nomophobia.
Smartphone Addiction Survey (Young Population) | through study completion, an average of 1 year
  The scale consists of 33 questions and 7 sub-parameters in total. Sub-parameters Functioning Impairment, Withdrawal Symptom, Positive Expectation, Virtual Directed Relationship, Overuse, Social Network Addiction, and Physical are symptoms. As the score increases, the level of addiction increases.

SECONDARY OUTCOMES:
Cervical Radiography | through study completion, an average of 1 year
  C2-7 Cobb Angle

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin ŞAHBAZ, Asis.Prof, Study Director — University Beykent
Locations (1):
- Yasemin ŞAHBAZ, Beylikduzu, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reed MD, Van Nostran W. Assessing pain intensity with the visual analog scale: a plea for uniformity. J Clin Pharmacol. 2014 Mar;54(3):241-4. doi: 10.1002/jcph.250. Epub 2014 Jan 23. No abstract available. PMID 24374753
- [Result] Kwon M, Lee JY, Won WY, Park JW, Min JA, Hahn C, Gu X, Choi JH, Kim DJ. Development and validation of a smartphone addiction scale (SAS). PLoS One. 2013;8(2):e56936. doi: 10.1371/journal.pone.0056936. Epub 2013 Feb 27. PMID 23468893
- [Result] Lee S, Kang H, Shin G. Head flexion angle while using a smartphone. Ergonomics. 2015;58(2):220-6. doi: 10.1080/00140139.2014.967311. Epub 2014 Oct 17. PMID 25323467
- [Result] Eitivipart AC, Viriyarojanakul S, Redhead L. Musculoskeletal disorder and pain associated with smartphone use: A systematic review of biomechanical evidence. Hong Kong Physiother J. 2018 Dec;38(2):77-90. doi: 10.1142/S1013702518300010. Epub 2018 Aug 14. PMID 30930581